CLINICAL TRIAL: NCT02789553
Title: Starches Digestion After Obesity Surgery. A Comparative Study.
Brief Title: Starches Digestion After Obesity Surgery.
Acronym: GLUBYPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 13 196 02; 2015-A01346-43 (Other: RCB)
Record Dates: First submitted 2016-03-24; First posted 2016-06-03 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Obesity
Keywords: Glucose digestion; Bypass surgery; C13-glucose tracer; Insulin secretion
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meal with glucose syrup (Experimental): Meal with glucose syrup : 30g of glucose mixed with 150 mL of water and dived into three 50 mL portions. It will be consumed in 15 minutes
  Interventions: Other: First starch meal then meal with glucose syrup; Other: First meal with glucose syrup then starch meal
- Starch meal (Experimental): Starch meal with 30g mixed in 120 mL of water. It will be consumed in 15 minutes and it represents 30g of glucose
  Interventions: Other: First starch meal then meal with glucose syrup; Other: First meal with glucose syrup then starch meal

INTERVENTIONS:
Other: First starch meal then meal with glucose syrup — Before bypass surgery, patients will take randomized meal. One day a starch meal and another day a glucose syrup meal. 3 months after surgery, they will take these 2 randomized meal again, one day the first one, and the day after the other one.
Other: First meal with glucose syrup then starch meal — Before bypass surgery, patients will take randomized meal. One day a meal with glucose syrup and another day a starch meal. 3 months after surgery, they will take these 2 randomized meal again, one day the first one, and the day after the other one.

SUMMARY:
Despite an impressive capacity to induce diabetes remissions, the gastric bypass surgery has been associated with the onset of hyperglycemic peaks, which are very intensive and transient, in formally non diabetic patients. The aim of this study is to study the digestion of starch as compared to that of glucose (same glucose load) before and after gastric bypass surgery in obese patients.

Volunteers will be recruited among the candidates to a gastric bypass, and will be studied before and 3 months after surgery. They will have on each occasion 2 random meals, corresponding to 30g glucose, one made of starch the other made of glucose, both naturally labeled with 13C. The digestion of starch will be assessed with the increase in the plasma 13C-glucose tracer. Plasma samples will be collected for 3 hours.

Some studies have already investigated time of absorption of glucose, but any study has examined the time of digestion of glucose. Other study always used glucose syrup, so they cannot have results about digestion. It is the reason why, in this study, glucose syrup and a starch meal will be taken by the same patient and glycaemia will be compared. In this way, results will be obtained about the kinetic of digestion of starch.

DETAILED DESCRIPTION:
Despite an impressive capacity to induce diabetes remissions, the gastric bypass surgery has been associated with the onset of hyperglycemic peaks, which are very intensive and transient, in formally non diabetic patients. The aim of this study is to study the digestion of starch as compared to that of glucose (same glucose load) before and after gastric bypass surgery in obese patients.

Volunteers will be recruited among the candidates to a gastric bypass, and will be studied before and 3 months after surgery. They will have on each occasion 2 random meals, corresponding to 30g glucose, one made of starch the other made of glucose, both naturally labeled with 13C. The digestion of starch will be assessed with the increase in the plasma 13C-glucose tracer. Plasma samples will be collected for 3 hours.

Some studies have already investigated time of absorption of glucose, but any study has examined the time of digestion of glucose. Other study always used glucose syrup, so they cannot have results about digestion. It is the reason why, in this study, glucose syrup and a starch meal will be taken by the same patient and glycaemia will be compared. In this way, results will be obtained about the kinetic of digestion of starch.

All patients will have two evaluations: one before the bypass surgery and one 3 months after. All evaluation will include 2 standard meals. Patients have to be fasted, and they will take in a randomized order the same glucose quantity: 30g, for the breakfast. After each meal, blood sample will be collected during 3 hours at time 0, 10, 20, 30, 40, 50, 60 minutes and every 30 minutes until time 180.

The starch meal will provide 30g of glucose in the form of corn starch. It will be consumed in 15 minutes. They are any other food in the meal. This quantity is corresponding to what patients can ingest after a bypass surgery, because of the poor size of their stomach. C13-carbon is a natural tracer into the corn. The measure of the increase of C13-glucose in the plasma is showing the appearance of the tracer, corresponding to the starch digestion.

The second meal is composed by 30g of corn glucose (glucose-meal), in liquid form and will be dived in 3 portions to be ingested in 15 minutes, like the starch meal. They are any other food in the meal.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients before obesity-surgery (HAS 2009 criteria for obesity-surgery)
* Patients accepted for a gastric bypass
* Patient consent the principle of 2 evaluations (one before surgery and another 3 months after surgery)
* Patient that give their informed consent before any procedure for the study
* Patient affiliated with a health insurance scheme

Exclusion Criteria:

* Diabetes (whatever the treatment), post-surgery diarrhea, small intestine disease
* Known microbial outbreak
* Anti-thrombin therapy
* Treatment which can modify the intestinal transit (anti-diarrhea, thyroid hormones…)
* Pregnant woman or breastfeeding.
* Patient not available for the two evaluations
* Protected adults (guardianship by court order)
* Patients participating to another treatment research protocol during the time of this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
Change in C13 glucose marker appearance: starch diet. | Change from baseline C13 glucose marker appearance at 3 months after surgery
  Appearance of the C13-glucose tracer in the plasma, since the beginning of the diet with the starch diet.

SECONDARY OUTCOMES:
C13 glucose marker appearance: glucose diet. | Change from baseline C13 glucose marker appearance at 3 months after surgery
  Appearance of the C13-glucose tracer in the plasma, since the beginning of the diet with the glucose diet.
Insulin secretion | Change from baseline insulin secretion at 3 months after surgery
  Insulin secretion will be measured with a deconvolution model.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick RITZ, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Department of Endocrinology, metabolic diseases and nutrition, Toulouse, France

IPD SHARING:
Plan to Share IPD: No